CLINICAL TRIAL: NCT02006992
Title: Growth of Infants Fed Hydrolysate Formulas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: AJ57
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Growth and Tolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RTF Infant Formula 1 (Active Comparator): a ready to feed (RTF) extensively hydrolyzed infant formula fed ad lib.
  Interventions: Other: RTF Infant Formula
- Powder Infant Formula 2 (Experimental): a powdered extensively hydrolyzed infant formula fed ad lib.
  Interventions: Other: Powder Infant Formula

INTERVENTIONS:
Other: RTF Infant Formula — a RTF extensively hydrolyzed infant formula
  Arms: RTF Infant Formula 1
Other: Powder Infant Formula — a powdered extensively hydrolyzed infant formula.
  Arms: Powder Infant Formula 2

SUMMARY:
Effects on weight and weight gain will be monitored in healthy term infants fed assigned infant formulas.

ELIGIBILITY:
Inclusion Criteria:

* Infants in good health.
* Singleton, term birth with a gestational age of 37 to 42 weeks.
* Birth weight of 2500 g (5 lb 8 oz) or greater.
* Between 0 and 9 days of age at enrollment.
* Not receiving vitamin or mineral supplements.

Exclusion Criteria:

- Maternal, fetal or perinatal medical history with potential for adverse effects on growth or development.

Max Age: 9 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 195 (Actual)
Dates: Start 2000-03; Primary Completion 2000-11 (Actual); Study Completion 2000-11 (Actual)

PRIMARY OUTCOMES:
Weight | Study day 1 to 112 days of age

SECONDARY OUTCOMES:
Length | Study day 1 to 112 days of age
Head Circumference | Study day 1 to 112 days of age
Study Formula Intake | Enrollment to 112 days of age
Incidence of Spit Up | Enrollment to 112 days of age
Stool Pattern | Enrollment to 112 days of age

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Borschel, RD, PhD, Study Chair — Abbott Nutrition
Locations (8):
- United States (8):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Dreyer Medical Center, Aurora, Illinois
  - PediaResearch, LLC, Evansville, Indiana
  - The University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Kentucky Pediatric Research, Bardstown, Kentucky
  - Children's Mercy Hospital, Kansas City, Missouri
  - NC Children's & Young Adults' Clinical Research Foundation, Chapel Hill, North Carolina
  - GrandView Medical Research, Sellersville, Pennsylvania